CLINICAL TRIAL: NCT05769088
Title: Effects of a Protein-Based Multi-Ingredient Pre-Workout Supplement on Body Composition, Performance, Perceptual Responses, Energy Feelings and Muscular Properties, in Middle-Aged and Older Adults.
Brief Title: Effects of a Multi-Ingredient Pre-Workout Supplement on Body Composition, Performance, Muscular Properties, and Wellbeing in Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Joel Puente (Other)
Collaborators: Crown Sport Nutrition (Industry); Go Fit Spain (Unknown)
Responsible Party: Sponsor-Investigator, Joel Puente, Principal Investigator, University of Greenwich
Organization: University of Greenwich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGreenwich3
Record Dates: First submitted 2023-02-20; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Protein Deficiency; Training Group, Sensitivity; Fatigue; Muscular Atrophy; Psychological
Keywords: Fatigue; Supplement; Protein; Resistance Training; Pre-workout; Strength; Rate of Perceived Exertion; Muscle
MeSH Terms: conditions — Protein Deficiency; Hypersensitivity; Fatigue; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: 6 Weeks of resistance training (alternate days), with a Pre-workout or Maltodextrin intake.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Ingredient Pre-Workout Supplement (Experimental): A 60 g dose of a commercially available preworkout supplement providing 159 kcal including carbohydrates 15 g, essential amino acids 12 g, citrulline 3.5 g, Arginine, 3.5 g Taurine 1 g, L-Tyrosine
  1 g, yerba mate 0.3 g and caffeine 0.4 g. With 350 ml of water.
  Interventions: Dietary Supplement: Ingestion of a Pre-Workout Supplement
- Maltodextrin Supplement (Placebo Comparator): A isoenergetic Maltodextrin supplement will be administered as placebo. With 350 ml of water.
  Interventions: Dietary Supplement: Ingestion of a Maltodextrin Supplement

INTERVENTIONS:
Dietary Supplement: Ingestion of a Pre-Workout Supplement — The Multi-Ingredient Pre-Workout Supplement is administered 15 minutes before the beginning of training sessions. No supplementation is administered in non-training days.
  The Resistance Training is performed in alternate days. The training Protocol is: 10 minutes of standardized warm-up, Strength Circuit training using free weights (Alternate Box Step-Ups, Bench Press; Parallel Squat; Up-right Row; Deadlift; Alternate Lunges; Shoulder Press; Leg Extension). The participants perform 16 repetitions of each exercise, with 30 seconds rest and 3 minutes rest after every set. If they can complete 16 repetitions easily, 2.5 to 5 kg are added for the next set. Also, whole-body Perceptual Response is assessed using the 0-10 OMNI-RES Scale, after every set and 15 minutes after finishing.
  Arms: Multi-Ingredient Pre-Workout Supplement
Dietary Supplement: Ingestion of a Maltodextrin Supplement — The Maltodextrin Supplement is administered 15 minutes before the beginning of training sessions. No supplementation is administered in non-training days.
  The Resistance Training is performed in alternate days. The training Protocol is: 10 minutes of standardized warm-up, Strength Circuit training using free weights (Alternate Box Step-Ups, Bench Press; Parallel Squat; Up-right Row; Deadlift; Alternate Lunges; Shoulder Press; Leg Extension). The participants perform 16 repetitions of each exercise, with 30 seconds rest and 3 minutes rest after every set. If they can complete 16 repetitions easily, 2.5 to 5 kg are added for the next set. Also, whole-body Perceptual Response is assessed using the 0-10 OMNI-RES Scale, after every set and 15 minutes after finishing.
  Arms: Maltodextrin Supplement

SUMMARY:
The investigation will be conducted as a double blinded, randomized, parallel between treatment conditions comparison design with two different groups ingesting a different supplement each one.

DETAILED DESCRIPTION:
Following inclusion, familiarization and baseline assessments, the participants will be randomly allocated to receive either a multi-ingredient, pre-workout supplement (PREW) or maltodextrin (CHO). Thereafter, the participants will follow a 6-weeks resistance training mesocycle, involving three resistance training sessions (Monday, Wednesday and Friday) per week (18 sessions in total). Before and after the 6 weeks of intervention, the following assessments will be performed: (i) Body composition (fat mass and fat-free mass) via air displacement plethysmography (BodPod); (ii) muscle contractile properties on Vastus Medialis and Anterior Deltoids (via Tensiomyography; (iii) muscle structure of the Vastus Lateralis of the Quadriceps and the Elbow Flexors of dominant extremities via Ultrasound; (iv) Maximal Isometric Strength (Isometric Mid-Thigh Pull); (v) Upper and Lower Body Muscular Power (Medicine Ball Throw and Vertical Jump), (vi) Upper and Lower Muscular Endurance (30-Seconds Sit-to-Stand and 30-Seconds 16RM Bench Press), (vii) Immune System (via HemoCue WBC DIFF System).

The supplements will be ingested 15 min before each training session.

Energy Feeling Questionnaire will be filled immediately before warming up.

In addition, Rate of Perceived Exertion to training will be assessed 15 min after the completion of all workouts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no injuries, illnesses or medication intake).
* Between 45 and 65 years old.
* Active and familiarised with Resistance Training.

Exclusion Criteria:

* Unhealthy (illnesses or medication intake) or injured.
* Untrained.
* Young (<45 y.o.) or elderly (>65 y.o.).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Tensiomyography | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  A TMG portable device (TMG Measurement System, 146 TMG-BMC Ltd., Ljubljana, Slovenia) with a maximal stimulation output of 110 mA·ms-1 IS used to evaluate the contractile properties of the Anterior Deltoid (AD) of the dominant limb. Changes in the evoked muscular contractile properties are estimated by analysing maximal radial displacement of the muscle belly in millimetres (Dm).
Vertical Jump | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  Height (measured in centimetres)
Chest Medicine Ball Throw | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  Medicine Ball Throw (measured in meters and centimetres).
Maximal Mid-Thigh Pull Isometric Strength | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  Maximal Strength (measured in kilograms).
Muscle Thickness | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  Thickness of the Vastus Lateralis and the Elbow Flexors of the dominant limbs
Self Perceived Energy Feeling | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  All participants will fill a short questionnaire (from 1 to 5 points) about their perception of energy before every training.
  Energy Feeling will be assessed (Evergy level, Fatigue Level, Feeling of Alertness, and Feeling of Focus for the task, valued from 1 = low energy to 5 = high energy).
Whole Body Perceptual Response during Resistance Training | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  Self Rate of Perceived Exertion (RPE) will be assessed via OMNI RES Scale (0-10 values) during resistance training (after every circuit) and 15-20 minutes after finishing each session.

SECONDARY OUTCOMES:
White Blood Cells count | Changes from 3 days previous to, and 3 days after the completion of the 6-weeks training program
  White blood cell (WBC) count including a five-part differential.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Greenwich, Avery Hill Campus, Sparrows Farm. Avery Hill, London., United Kingdom, SE9 2BT, London, Avery Hill, London., United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puente-Fernandez J, Larumbe-Zabala E, Roberts J, Naclerio F. Effect of a Multi-Ingredient Post-Workout Dietary Supplement on Body Composition and Muscle Strength - A Randomized Controlled Trial. J Diet Suppl. 2025;22(3):445-462. doi: 10.1080/19390211.2025.2488811. Epub 2025 Apr 12. PMID 40219860